CLINICAL TRIAL: NCT03167606
Title: A Pragmatic Clinical Trial of MyPEEPS Mobile to Improve HIV Prevention Behaviors in Diverse Adolescent MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Washington (Other); New York Blood Center (Other); University of Alabama at Birmingham (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Assistant Professor of Disease Prevention and Health Promotion in the Faculty of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAQ6500; U01MD011279 (NIH)
Record Dates: First submitted 2017-05-11; First posted 2017-05-30 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: HIV Infections
Keywords: myPEEPS; Mobile Intervention; Human Immunodeficiency Virus (HIV); Men who have sex with men (MSM)
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Study participants randomized to the immediate intervention arm will have access to the MyPEEPS Mobile from the baseline visit to 3-month follow-up visit. They will continue with follow-up visits at 6 months and 9 months, but will no longer have access to the MyPEEPS Mobile past the 3-month follow-up visit.
  Interventions: Behavioral: MyPEEPS Mobile
- Delayed Intervention (Experimental): Study participants randomized to the delayed intervention arm will complete visits at baseline, 3 months, 6 months, 9 months, and 12 months. They will have access to the MyPEEPS Mobile from the 9-month follow-up visit until the 12-month follow-up visit.
  Interventions: Behavioral: MyPEEPS Mobile

INTERVENTIONS:
Behavioral: MyPEEPS Mobile — Mobile technology to deliver HIV prevention information specifically developed for at-risk YMSM.

SUMMARY:
The proposed MyPEEPS Mobile intervention is a novel and evidence-driven intervention using mobile technology to deliver HIV prevention information specifically developed for at-risk young men who have sex with men (YMSM). This will be the one of the first studies to test the efficacy of a scaled-up, mobile version of an existing human immunodeficiency virus (HIV) prevention intervention originally developed for, designed by, and piloted for, a diverse group of YMSM.

MyPEEPS Mobile will be tested in an randomized controlled trial with racially and ethnically diverse HIV-negative or unknown status YMSM aged 13-18 at four geographically diverse sites: Birmingham, Chicago, New York City, and Seattle, allowing for increased generalizability of findings.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) bear a greater burden of HIV/AIDS than any other population group in the US, comprising only 2% of the population but 56% of individuals living with HIV/AIDS. Although much of the increased incidence in HIV has been reported among YMSM, especially among racial and ethnic minority groups, and is linked to high-risk sexual behavior, there remains a dearth of evidence-based HIV prevention interventions for YMSM - and none that address racially/ethnically diverse YMSM. To address this need, this study leverages mobile technology and MyPEEPS, an existing theory-driven, multi-ethnic, group-level, evidence-based intervention for diverse YMSM. MyPEEPS is a manualized curriculum, comprised of 6 modules focusing on key intermediate social and personal factors, including knowledge (e.g., correct way to use a condom), self-efficacy for safer sex, interpersonal communication skills and behavioral skills. MyPEEPS is one of the only HIV prevention interventions in the literature that focuses on diverse adolescent MSM. Long-term sustainability of face-to face, group-level behavioral interventions, such as MyPEEPS, have been problematic for dissemination in at-risk populations, particularly among young racial and ethnic minority groups. In response to this challenge, the investigators propose to translate MyPEEPS from a face-to-face, group-based curriculum to a mobile, responsive-driven web-based platform, accessible by smartphone or other web-enabled devices, to increase accessibility and scalability for diverse YMSM. The ubiquitous nature of mobile phones in daily life, especially among 13-18 year olds, has created opportunities for health interventions in a portable format with enhanced privacy. Using a participatory approach, this study will incorporate user-centered design in the translation of the MyPEEPS intervention onto a mobile platform.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as male, nonbinary, or genderqueer
* Male sex assigned at birth
* Understand and read English
* Live in the United States or its territories
* Own or have access to a mobile device (e.g., smartphone or tablet)
* Same-sex attraction and either kissed another guy or intending to engage in sexual activity with another guy in next year
* Self-report HIV-negative or unknown status

Exclusion Criteria:

* HIV+

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants must identify as male, nonbinary, or genderqueer
Enrollment: 764 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, Principal Investigator — Columbia University School of Nursing
Locations (4):
- United States (4):
  - Birmingham Aids Outreach, Birmingham, Alabama
  - Lurie Children's Hospital, Chicago, Illinois
  - Columbia University School of Nursing, New York, New York
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cordoba E, Garofalo R, Kuhns LM, Pearson CR, Batey DS, Bruce J, Radix A, Belkind U, Hidalgo MA, Hirshfield S, Schnall R. A Cross-sectional Study of Perceived Stress and Racial Discrimination Among a National Sample of Young Men Who Have Sex With Men. J Assoc Nurses AIDS Care. 2023 May-Jun 01;34(3):226-237. doi: 10.1097/JNC.0000000000000407. PMID 37129475
- [Derived] Schnall R, Kuhns LM, Pearson C, Batey DS, Bruce J, Hidalgo MA, Hirshfield S, Janulis P, Jia H, Radix A, Belkind U, Rodriguez RG, Garofalo R. Efficacy of MyPEEPS Mobile, an HIV Prevention Intervention Using Mobile Technology, on Reducing Sexual Risk Among Same-Sex Attracted Adolescent Males: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2231853. doi: 10.1001/jamanetworkopen.2022.31853. PMID 36129712
- [Derived] Diaz JE, Sandh S, Schnall R, Garofalo R, Kuhns LM, Pearson CR, Bruce J, Batey DS, Radix A, Belkind U, Hidalgo MA, Hirshfield S. Predictors of Past-Year Health Care Utilization Among Young Men Who Have Sex with Men Using Andersen's Behavioral Model of Health Service Use. LGBT Health. 2022 Oct;9(7):471-478. doi: 10.1089/lgbt.2021.0488. Epub 2022 Jul 22. PMID 35867076
- [Derived] Cordoba E, Kuizon CM, Garofalo R, Kuhns LM, Pearson C, Batey DS, Bruce J, Radix A, Belkind U, Hidalgo MA, Hirshfield S, Jia H, Schnall R. Are State-Level HIV Testing Policies for Minors Associated With HIV Testing Behavior and Awareness of Home-Based HIV Testing in Young Men Who Have Sex With Men? J Adolesc Health. 2022 Jun;70(6):902-909. doi: 10.1016/j.jadohealth.2021.12.023. Epub 2022 Feb 28. PMID 35241362
- [Derived] Cordoba E, Garofalo R, Kuhns LM, Pearson C, Bruce J, Batey DS, Radix A, Belkind U, Hidalgo MA, Hirshfield S, Garibay Rodriguez R, Schnall R. Risk-taking behaviors in adolescent men who have sex with men (MSM): An association between homophobic victimization and alcohol consumption. PLoS One. 2021 Dec 2;16(12):e0260083. doi: 10.1371/journal.pone.0260083. eCollection 2021. PMID 34855787
- [Derived] Kuhns LM, Garofalo R, Hidalgo M, Hirshfield S, Pearson C, Bruce J, Batey DS, Radix A, Belkind U, Jia H, Schnall R. A randomized controlled efficacy trial of an mHealth HIV prevention intervention for sexual minority young men: MyPEEPS mobile study protocol. BMC Public Health. 2020 Jan 15;20(1):65. doi: 10.1186/s12889-020-8180-4. PMID 31941475

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled in error (ineligible age) and withdrawn from the study prior to randomization
Groups:
- Immediate Intervention: Study participants randomized to the immediate intervention arm will have access to the MyPEEPS Mobile from the baseline visit to 3-month follow-up visit. They will continue with follow-up visits at 6 months and 9 months, but will no longer have access to the MyPEEPS Mobile past the 3-month follow-up visit.
  MyPEEPS Mobile: Mobile technology to deliver HIV prevention information specifically developed for at-risk young men who have sex with men (YMSM).
Period: Overall Study
Arm/Group | Immediate Intervention | Delayed Intervention
Started | 382 | 381
Completed | 303 | 310
Not Completed | 79 | 71
Not completed — Lost to Follow-up | 73 | 64
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Withdrawal by Investigator | 0 | 2

BASELINE CHARACTERISTICS:
Population: The analytic sample included 760 of the 764 participants enrolled because 1 participant was enrolled in error (ineligible age) and withdrawn from the study prior to randomization and 3 participants were excluded from the analytic sample due to missing or invalid data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Delayed Intervention | Total
Number analyzed (Participants) | 379 | 381 | 760
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.23 (1.4) | 16.20 (1.4) | 16.22 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 379 | 381 | 760
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 169 | 142 | 311
  Not Hispanic or Latino | 210 | 239 | 449
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 23 | 43
  Asian | 36 | 36 | 72
  Native Hawaiian or Other Pacific Islander | 6 | 5 | 11
  Black or African American | 75 | 83 | 158
  White | 132 | 152 | 284
  More than one race | 55 | 39 | 94
  Unknown or Not Reported | 55 | 43 | 98
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 379 | 381 | 760
Any Anal Sex Acts With Another Male [Count of Participants; unit: Participants] | 203 | 192 | 395

OUTCOME MEASURES:

1. Primary Outcome: Number of Condomless Anal Sex Acts
Description: The number of condomless anal sex acts (CASA) will be evaluated at all time points using the AIDS-Risk Behavior Assessment (ARBA) adapted for YMSM. At each timepoint, participants were asked to report the past 3 month number of insertive and receptive anal sex acts during which condoms were not used.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: condomless anal sex acts
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
condomless anal sex acts
  Baseline | 1.53 (0.29) | 1.45 (0.27)
  3-Month Follow-up | 1.04 (0.26) | 1.63 (0.38)
  6-Month Follow-up | 1.68 (0.47) | 1.21 (0.25)
  9-Month Follow-up | 1.70 (0.36) | 1.65 (0.33)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 1.47 (0.36)

2. Primary Outcome: Number of Anal Sex Partners
Description: The number of anal sex partners will be evaluated at all time points using the AIDS-Risk Behavior Assessment (ARBA) adapted for YMSM. Participants are asked to report the number of insertive and receptive anal sex partners in their lifetime at the baseline timepoint and then asked to report the number of insertive and receptive anal sex partners in the past 3 months at each of the follow-up timepoints.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Anal sex partners
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
Anal sex partners
  Baseline | 0.95 (0.11) | 0.87 (0.09)
  3-Month Follow-up | 0.86 (0.13) | 0.71 (0.09)
  6-Month Follow-up | 0.90 (0.11) | 0.84 (0.10)
  9-Month Follow-up | 1.00 (0.13) | 0.77 (0.08)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 1.27 (0.21)

3. Primary Outcome: Number of Condomless Anal Sex Partners
Description: The number of condomless anal sex (CAS) partners will be evaluated at all time points using the AIDS-Risk Behavior Assessment (ARBA) adapted for YMSM. Participants are asked to report the number of insertive and receptive anal sex partners with whom condoms were not used in their lifetime at the baseline timepoint and then asked to report the number of insertive and receptive anal sex partners with whom condoms were not used in the past 3 months at each of the follow-up timepoints.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Condomless anal sex partners
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
Condomless anal sex partners
  Baseline | 0.53 (0.08) | 0.42 (0.05)
  3-Month Follow-up | 0.50 (0.08) | 0.38 (0.06)
  6-Month Follow-up | 0.43 (0.06) | 0.47 (0.06)
  9-Month Follow-up | 0.63 (0.11) | 0.40 (0.05)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 0.72 (0.17)

4. Primary Outcome: Number of Anal Sex Acts Under the Influence of Drugs/Alcohol
Description: The number of anal sex acts under the influence of drugs/alcohol will be evaluated at all time points using the AIDS-Risk Behavior Assessment (ARBA) adapted for YMSM. At each timepoint, participants were asked to report the past 3 month number of insertive and receptive anal sex acts during which they had been drinking alcohol or using drugs.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Anal sex acts under the influence
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
Anal sex acts under the influence
  Baseline | 0.33 (0.09) | 0.45 (0.11)
  3-Month Follow-up | 0.35 (0.16) | 0.42 (0.14)
  6-Month Follow-up | 0.35 (0.18) | 0.43 (0.09)
  9-Month Follow-up | 0.41 (0.11) | 0.54 (0.12)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 0.53 (0.16)

5. Primary Outcome: Number of Participants With Self-reported Pre-exposure Prophylaxis (PrEP) Use
Description: Participants were asked if they have ever used Pre-exposure Prophylaxis (PrEP) at baseline, if they have used PrEP in the prior 3 months at all timepoints, and if they are currently using PrEP at the time of study visit at all timepoints.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
Participants
  Baseline | 10 | 10
  3-Month Follow-up: number analyzed (Participants) | 320 | 338
  3-Month Follow-up | 14 | 14
  6-Month Follow-up: number analyzed (Participants) | 304 | 321
  6-Month Follow-up | 20 | 16
  9-Month Follow-up: number analyzed (Participants) | 306 | 317
  9-Month Follow-up | 13 | 14
  12-Month Follow-up: number analyzed (Participants) | 0 | 309
  12-Month Follow-up |  | 25

6. Primary Outcome: Number of Participants With Self-reported Non-occupational Post-Exposure Prophylaxis (nPEP) Use
Description: Participants were asked if they've ever used Non-occupational Post-Exposure Prophylaxis (nPEP) at baseline and if they've used nPEP in the 3 months prior to each study visit timepoint.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
Participants
  Baseline | 4 | 6
  3-Month Follow-up: number analyzed (Participants) | 320 | 338
  3-Month Follow-up | 3 | 4
  6-Month Follow-up: number analyzed (Participants) | 304 | 321
  6-Month Follow-up | 5 | 8
  9-Month Follow-up: number analyzed (Participants) | 306 | 317
  9-Month Follow-up | 1 | 3
  12-Month Follow-up: number analyzed (Participants) | 0 | 309
  12-Month Follow-up |  | 3

7. Primary Outcome: Number of Participants With Self-Reported HIV Testing
Description: Participants were asked to report how many times they've ever been tested for HIV at baseline and at each follow-up timepoint they were asked how many times they've tested for HIV in the prior 3 months.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
Participants
  Baseline | 63 | 55
  3-Month Follow-up: number analyzed (Participants) | 320 | 338
  3-Month Follow-up | 90 | 79
  6-Month Follow-up: number analyzed (Participants) | 304 | 321
  6-Month Follow-up | 84 | 69
  9-Month Follow-up: number analyzed (Participants) | 306 | 317
  9-Month Follow-up | 93 | 69
  12-Month Follow-up: number analyzed (Participants) | 0 | 309
  12-Month Follow-up |  | 71

8. Primary Outcome: Number of Participants With Self-Reported Sexually Transmitted Infection (STI) Testing
Description: Participants were asked to report past 3-month testing for sexually transmitted infections (STIs) at each timepoint.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
Participants
  Baseline | 73 | 65
  3-Month Follow-up: number analyzed (Participants) | 320 | 338
  3-Month Follow-up | 63 | 49
  6-Month Follow-up: number analyzed (Participants) | 304 | 321
  6-Month Follow-up | 56 | 44
  9-Month Follow-up: number analyzed (Participants) | 306 | 317
  9-Month Follow-up | 59 | 44
  12-Month Follow-up: number analyzed (Participants) | 0 | 309
  12-Month Follow-up |  | 53

9. Secondary Outcome: Intent to Have Anal Sex
Description: Participants were presented with the statement "During the next 3 months, I am not planning to have anal sex" with response options ranging from 1=Very true to 4=Very untrue. The mean value was calculated per group and per timepoint.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
score on a scale
  Baseline | 2.35 (0.06) | 2.40 (0.05)
  3-Month Follow-up | 2.30 (0.06) | 2.36 (0.06)
  6-Month Follow-up | 2.33 (0.06) | 2.35 (0.06)
  9-Month Follow-up | 2.42 (0.06) | 2.40 (0.06)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 2.42 (0.06)

10. Secondary Outcome: Intent to Always Use Condoms During Anal Sex With All Sex Partners
Description: Participants responded to the statement "During the next 3 months, I plan to always use condoms during anal sex with all of my sex partners" with response options ranging from 1=Very true to 4=Very untrue. Mean values were calculated by group for each timepoint.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
units on a scale
  Baseline | 3.38 (0.04) | 3.41 (0.04)
  3-Month Follow-up | 3.45 (0.05) | 3.44 (0.04)
  6-Month Follow-up | 3.34 (0.05) | 3.37 (0.05)
  9-Month Follow-up | 3.42 (0.05) | 3.38 (0.04)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 3.35 (0.05)

11. Secondary Outcome: Intent to Use PrEP as a Strategy to Reduce HIV Infection Risk
Description: Participants responded to the statement "I plan to use PrEP as a strategy to reduce my risk for HIV infection during the next three months" with response values ranging from 1=Very true to 4=Very untrue. Mean values were calculated for each group at each timepoint.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
units on a scale
  Baseline | 2.67 (0.06) | 2.65 (0.05)
  3-Month Follow-up | 2.82 (0.06) | 2.66 (0.06)
  6-Month Follow-up | 2.79 (0.06) | 2.66 (0.06)
  9-Month Follow-up | 2.74 (0.06) | 2.59 (0.05)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 2.83 (0.06)

12. Other Pre Specified Outcome: Self-efficacy for Safer Sex and Situational Temptation for Unsafe Sex
Description: Participants were asked to respond to 10 questions assessing self-efficacy in practicing condom use and safer sex communication with a partner. A sample item is "if I didn't want to have sex with my partner, I would be able to say no." Response options ranged from 1=Strongly agree to 4=Strongly disagree. Question scores ranged 1-4, values averaged and total scores ranged from 1 to 4, with lower values indicating higher self-efficacy
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
units on a scale
  Baseline | 1.51 (0.02) | 1.52 (0.02)
  3-Month Follow-up | 1.44 (0.02) | 1.54 (0.02)
  6-Month Follow-up | 1.50 (0.02) | 1.52 (0.02)
  9-Month Follow-up | 1.47 (0.02) | 1.55 (0.02)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 1.44 (0.02)

13. Other Pre Specified Outcome: Condom Use Errors
Description: The condom errors survey is a 12-item questionnaire was adapted to reflect a 6-week recall period. A sample question is "when you used condoms during the last six weeks, how often was the condom put on the wrong side up so that it had to be flipped over?" Response options ranged from 0=Never to 2=Always. Question scores ranged 0-2, values averaged and total scores ranged from 0 to 2, with lower values indicating fewer condom use errors.
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Intervention | Delayed Intervention
Number analyzed (Participants) | 379 | 381
units on a scale
  Baseline | 0.60 (0.01) | 0.61 (0.01)
  3-Month Follow-up | 0.68 (0.01) | 0.59 (0.01)
  6-Month Follow-up | 0.67 (0.01) | 0.58 (0.01)
  9-Month Follow-up | 0.62 (0.01) | 0.57 (0.01)
  12-Month Follow-up: number analyzed (Participants) | 0 | 381
  12-Month Follow-up |  | 0.64 (0.02)

ADVERSE EVENTS:
Time Frame: Baseline, 3, 6, and 9 months (Intervention group); Baseline, 3, 6, 9, and 12 months (Delayed Intervention group)
Arm/Group | Immediate Intervention | Delayed Intervention
All-Cause Mortality (participants affected / at risk) | 0/382 | 0/381
Serious Adverse Events (participants affected / at risk) | 0/382 | 0/381
Other Adverse Events (participants affected / at risk) | 0/382 | 0/381

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT03167606/Prot_SAP_000.pdf